CLINICAL TRIAL: NCT04478890
Title: Hemodynamic Assessment of the Right Ventricle Using Pressure-volume Loop Catheter and Pulmonary Artery Catheter in Patients Undergoing Left Ventricular Assist Device Placement at the University of Minnesota Medical Center
Brief Title: Hemodynamic Assessment of the Right Ventricle Using Pressure-volume Loop Catheter and Pulmonary Artery Catheter in Patients Undergoing Left Ventricular Assist Device Placement
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: ANES-2020-28725
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Characterize right ventricular function while undergoing LVAD implantation
  Interventions: Diagnostic Test: Hemodynamic assessment

INTERVENTIONS:
Diagnostic Test: Hemodynamic assessment — Hemodynamic assessment of the right ventricle using pressure-volume loop catheter and pulmonary artery catheter

SUMMARY:
This study will include the placement of a pressure volume (PV) loop catheter in the right atrium of patients undergoing left ventricular assist device (LVAD) placement and measure relevant PV loop data. Transesophageal echocardiography (TEE) and pulmonary artery (PA) catheter parameters as comparators to the PV loop will be recorded.

DETAILED DESCRIPTION:
This will be a prospective observational study design to characterize right ventricular function in 5 consecutive patients undergoing LVAD implantation at the University of Minnesota Medical Center (UMMC). Pre-, intra- and postoperative care delivery to all enrolled and consented patients will meet the standards of care otherwise delivered to patients undergoing LVAD implantation at UMMC; care delivery will be at the discretion of the clinical care team and will not be altered based on the output of the right ventricular high-fidelity conductance catheters.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergoing left ventricular assist device (LVAD) placement at the University of Minnesota Medical Center

Exclusion Criteria:

* Patients with a history of internal jugular vein thrombosis or known reasons for not being able to thread a central venous catheter through either internal jugular vein
* Patients with a history of known esophageal strictures, esophageal or stomach cancer, esophageal varices, or any patient in whom a TEE is contraindicated
* Patients with permanent pacemakers whose right ventricle is being paced and not in normal sinus rhythm
* Patients unable to consent to participating in the study
* Patients who are pregnant will be excluded, as part of standard care, all female patients are screened for pregnancy prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients 18 years or older undergoing left ventricular assist device (LVAD) placement at the University of Minnesota Medical Center
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stroke volume | Approximately 4-6 hours
  Stroke volume will be reported in units of millilitres per square metre
Heart rate | Approximately 4-6 hours
  Heart rate will be reported in units of beats per minute
Ejection fraction | Approximately 4-6 hours
  Ejection fraction will be reported as a percent
Cardiac output | Approximately 4-6 hours
  Cardiac output will be reported in units of milliliters per minute
End-systolic pressure | Approximately 4-6 hours
  End-systolic pressure will be reported in units of mmHG
End-systolic volume | Approximately 4-6 hours
  End-systolic volume will be reported in units of milliliters
End-diastolic pressure | Approximately 4-6 hours
  End-diastolic pressure will be reported in units of mmHG
End-diastolic volume | Approximately 4-6 hours
  End-diastolic volume will be reported in units of milliliters
Right ventricular dP/dt | Approximately 4-6 hours
  Right ventricular dP/dt will be reported in units of mmHg per second
Stroke work | Approximately 4-6 hours
  Stroke work will be reported in units of gram meters (g*m)

CONTACTS AND LOCATIONS:
Overall Officials: Tjorvi Perry, MD, MMSc, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States